CLINICAL TRIAL: NCT00282217
Title: Sirolimus in the Treatment of Histological Defined Chronic Allograft Nephropathy
Brief Title: Study Evaluating Sirolimus in the Treatment of Kidney Transplant
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101467
Record Dates: First submitted 2006-01-24; First posted 2006-01-25 (Estimated); Last update posted 2007-03-22 (Estimated); Status verified 2007-03

CONDITIONS: Kidney Failure; Kidney Diseases
Keywords: Kidney Failure; Kidney Transplant; Graft Rejection; Kidney Transplantation
MeSH Terms: conditions — Renal Insufficiency; Kidney Diseases | interventions — Sirolimus

INTERVENTIONS:
Drug: Sirolimus

SUMMARY:
The aim of this study is to test whether withdrawal of calcineurin inhibitors, followed by treatment with sirolimus, may improve renal function in renal transplant recipients with chronic allograft nephropathy.

ELIGIBILITY:
Inclusion Criteria:

* Renal transplantation
* Biopsy-confirmed chronic rejection
* Treatment with mofetil mycophenolate among cyclosporine or tacrolimus

Exclusion Criteria:

* Transplant of any organ other than the kidney
* Current important infection
* Acute rejection within 12 weeks prior to inclusion

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2006-08

PRIMARY OUTCOMES:
Renal function at 12 months; Comparison between slopes of glomerular filtration rate (GFR) of one year before versus one year after start on sirolimus

SECONDARY OUTCOMES:
Histological parameters at 12 months
Cumulative incidence of biopsy-confirmed acute rejection at 12 months
Effect at 12 months on proteinuria, blood pressure, hyperlipidemia, and proteinuria

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Spain, infomed@wyeth.com
Locations (11):
- Spain (11):
  - A Coruña
  - Albacete
  - Barcelona
  - Cadiz
  - Granada
  - L'Hospitalet de Llobregat
  - Madrid
  - Málaga
  - Oviedo
  - Seville
  - Zaragoza